CLINICAL TRIAL: NCT02723188
Title: Modulation of Fear Extinction Processes Using Transcranial Electrical Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor of Psychology, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TASMC-13-TH-334
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Stress Related Disorder; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sham (Sham Comparator): Sham electrical stimulation
  Interventions: Device: Sham stimulation (1.5 milliampere,30 seconds)
- DC: Direct current (Experimental): Direct current electrical stimulation
  Interventions: Device: DC stimulation (1.5 milliampere, 20 minutes)
- AC: Alternating current (Experimental): Alternating current electrical stimulation
  Interventions: Device: AC stimulation (1.5 milliampere,1.5 Hertz frequency)

INTERVENTIONS:
Device: Sham stimulation (1.5 milliampere,30 seconds)
  Other Names: DC Stimulator Plus (neuroConn, Germany), serial 0118
  Arms: Sham
Device: DC stimulation (1.5 milliampere, 20 minutes)
  Other Names: DC Stimulator Plus (neuroConn, Germany), serial 0118
  Arms: DC: Direct current
Device: AC stimulation (1.5 milliampere,1.5 Hertz frequency)
  Other Names: DC Stimulator Plus (neuroConn, Germany), serial 0118
  Arms: AC: Alternating current

SUMMARY:
The aim of this study is to examine the effects of transcranial electrical stimulation on processes associated with fear extinction in healthy humans.

DETAILED DESCRIPTION:
Research links the processes of fear conditioning and extinction to the treatment of anxiety and stress-related disorders. Moreover, considerable translational research examines the neural correlates of these processes. However, virtually no research in humans manipulates neural correlates of these processes, which limits basic-clinical integration. The present study aimed to use transcranial electrical stimulation (tES) to modulate processes associated with fear extinction in order to assess the potential utility of tES in enhancing exposure-based treatment. To this end, healthy participants underwent a three-day fear conditioning and extinction paradigm. Participants were randomly assigned into 3 groups, differing in terms of tES applied during the extinction learning phase (Day 2) and targeting the medial prefrontal cortex: 1) direct current (DC) stimulation, aimed at enhancing extinction learning; 2) alternate current (AC) stimulation, aimed at interfering with reconsolidation of the fear memory activated during the extinction phase; and 3) sham stimulation. The outcome measures (outlined next) involve the assessment of extinction recall during a test phase (Day 3). Successful modulation of extinction learning by tES would be reflected in enhanced extinction recall.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* Self-reported major psychiatric condition
* Screening specific for electrical stimulation (psychotropic medication, metal implants in head, epilepsy or seizure history)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abend R, Jalon I, Gurevitch G, Sar-El R, Shechner T, Pine DS, Hendler T, Bar-Haim Y. Modulation of fear extinction processes using transcranial electrical stimulation. Transl Psychiatry. 2016 Oct 11;6(10):e913. doi: 10.1038/tp.2016.197. PMID 27727241

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham: Sham electrical stimulation
  Sham stimulation (1.5 milliampere,30 seconds)
- DC (Direct Current): Direct current electrical stimulation
  DC stimulation (1.5 milliampere, 20 minutes)
- AC (Alternating Current): Alternating current electrical stimulation
  AC stimulation (1.5 milliampere,1.5 Hertz frequency)
Period: Overall Study
Arm/Group | Sham | DC (Direct Current) | AC (Alternating Current)
Started | 15 | 15 | 15
Completed | 14 | 15 | 15
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DC: Direct Current: Direct current electrical stimulation
  DC stimulation (1.5 milliampere, 20 minutes)
- AC: Alternating Current: Alternating current electrical stimulation
  AC stimulation (1.5 milliampere,1.5 Hertz frequency)
- Total: Total of all reporting groups
Arm/Group | Sham | DC: Direct Current | AC: Alternating Current | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 45
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (7) | 23 (3) | 25 (5) | 25 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 8 | 22
  Male | 10 | 6 | 7 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  Israel | 15 | 15 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Galvanic Skin Response (GSR)
Description: GSR was measured throughout the task using 2 standard electrodes on the fingers. Measurement units were in micro-Siemens; scores were square-root-transformed (a common method in GSR studies). A higher level of GSR in response to stimuli is taken to reflect greater physiological fear response, and thus worse in the context of the relevance of the study conditions to the treatment of anxiety disorders.
  Scores were collected in response to presentation of the CS+ (the stimulus conditioned to be associated with an aversive outcome) and the CS- (the stimulus not conditioned to be associated with any outcome).
Time Frame: During three-day experimental task
Measure: Mean (Standard Deviation); unit: micro-Siemens
Arm/Group | Sham | DC: Direct Current | AC: Alternating Current
Number analyzed (Participants) | 14 | 15 | 15
micro-Siemens
  CS (conditioned stimulus)+ | .45 (.38) | .56 (.57) | .65 (.46)
  CS- | .23 (.25) | .54 (.54) | .24 (.38)

2. Secondary Outcome: Self-reported Fear Rankings
Description: Participants marked how fearful they are of stimuli used in the task on a single 10-point scale (1=not afraid, 10=extremely afraid). Higher scores therefore reflect greater fear and are worse in the context of treatment for anxiety disorders.
  Scores were collected in response to presentation of the CS+ (the stimulus conditioned to be associated with an aversive outcome) and the CS- (the stimulus not conditioned to be associated with any outcome).
Time Frame: During three-day experimental task
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham | DC: Direct Current | AC: Alternating Current
Number analyzed (Participants) | 14 | 15 | 15
units on a scale
  CS+ | 3.8 (2.5) | 4.7 (2.1) | 5.3 (2.5)
  CS- | 3.2 (2.0) | 2.5 (1.2) | 2.7 (2.2)

ADVERSE EVENTS:
Arm/Group | Sham | DC: Direct Current | AC: Alternating Current
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No